CLINICAL TRIAL: NCT02979002
Title: Accuracy of a Rapid Diagnostic Test for Cutaneous Leishmaniasis in Morocco
Status: Completed | Type: Observational
Sponsor: National School of Public Health, Morocco (Other)
Collaborators: Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Principal Investigator, Issam Bennis, MD, Doctor, National School of Public Health, Morocco
Other Study IDs: ENSP276/DGDB26012016
Record Dates: First submitted 2016-11-29; First posted 2016-12-01 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Cutaneous Leishmaniasis; Skin Diseases, Parasitic; Neglected Diseases
MeSH Terms: conditions — Leishmaniasis, Cutaneous; Skin Diseases, Parasitic; Neglected Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Suspected Cutaneous leishmaniasis lesions
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to estimate the accuracy of CL Detect Rapid Test™ compared to a composite reference standard test (Direct examination of skin smears + PCR test) in patients with clinically suspected Cutaneous Leishmaniasis disease in Morocco.

DETAILED DESCRIPTION:
Study participants are recruited in nine health centers located in fourthree CL endemic provinces. The RDT under evaluation (index test) is the CL Detect™ Rapid Test (InBios, USA); a membrane-based amastigote antigen (peroxidoxin) detection test. The reference standard consists of two tests: direct examination of skin smears and PCR. For each patient, the health professional takes one dental broach sample and four skin smear samples from a single lesion. The dental broach sample is used for the RDT, which is done once. The skin smear samples are sent to provincial laboratories for microscopy testing and to reference laboratories in Morocco and Belgium for PCR testing by ITS1 PCR, Hsp70 genotyping and parasite load determination. Readers of index and reference tests do not have access to clinical information or any other test results. The results of the test under evaluation (RDT) and the molecular tests (PCR) are not communicated to the patient or her/his physician, as case management has to follow current clinical guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Participants with suspected Cutaneous Leishmaniasis wound(s) in apparently healthy state
* Who is able to learn the Information sheet and sign the Informed consent form by them selves or by their parents with the presence or not of a witness (for illiterate people)
* Who satisfy the following criteria :

  * with an ulcerative lesion in any accessible part of the body to perform the dental broach and the scraping.
  * Just one ulcerative lesion by patient could be selected (The newest and the less infected)
  * Lesion should be less than 04 months of age

Exclusion Criteria:

* Patients with only nodular, papular, macular or nodulo-papular suspected CL forms
* Patients with ulcerative lesions with a suspected bacteria origin which could disappear after a short course of antibiotic treatment.
* Patients who already received during the last two months, prior to signing the consent, a physical treatment (e.g. cryotherapy, thermotherapy, Laser) or a traditional treatment (e.g. burn, acide, traditional scraping)
* Patients presenting other disease with the need to take anti-parasite treatments
* Patient with a acute or chronic disease needing hospitalization
* Patient who already received antimoniate treatment incomplete or complete duration and dose against CL
* Any situation that could engage the security of the patient or of the health professional (e.g. People with a psychiatric trouble or a mental handicap )
* For children less than 12 years old, the decision of participation is mainly based on the condition that their parents are able to learn and understand the information sheet and sign the informed consent form

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Primary health centers in Morocco
Sampling Method: Non-Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2016-12; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Positive result for this test | 50 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Issam Bennis, MD, MPH, Principal Investigator — National School of Public Health - Rabat - Morocco
Locations (9):
- Morocco (9):
  - Primary Health center, Arfoud, Errachidia
  - Health primary center, Tinajdad, Errachidia
  - Primary Health Center, Sekoura, Ouarzazates
  - Primary Health Center, Tarmight, Ouarzazates
  - Primary Health Center, Tazouta, Sefrou
  - Primary Health Center, Boumalne Dades, Tinghir
  - Primary Health Center, Kelaat Mgouna, Tinghir
  - Primary Health Center, Sefrou
  - Primary Health Center, Sidi Kacem

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bennis I, Verdonck K, El Khalfaoui N, Riyad M, Fellah H, Dujardin JC, Sahibi H, Bouhout S, Van der Auwera G, Boelaert M. Accuracy of a Rapid Diagnostic Test Based on Antigen Detection for the Diagnosis of Cutaneous Leishmaniasis in Patients with Suggestive Skin Lesions in Morocco. Am J Trop Med Hyg. 2018 Sep;99(3):716-722. doi: 10.4269/ajtmh.18-0066. Epub 2018 Jul 5. PMID 29988004